CLINICAL TRIAL: NCT01972932
Title: Protocol CHUM 2014-5056: A Randomized, Double Blinded Placebo Controlled Study to Evaluate the Efficacy of Bio-K+® in the Reduction of the Risk of Clostridium Difficile Infection and Antibiotic Associated Diarrhea in Hospitalized Patients
Brief Title: Study of Bio-K+® in the Reduction of the Risk of Clostridium Difficile Infection and Antibiotic Associated Diarrhea
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Bio-K Plus International Inc. (Industry)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHUM 2014-5056
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Clostridium Difficile Infection; Antibiotic Associated Diarrhea
Keywords: Bio-K+®; Placebo; AAD; CDI; hospitalized subjects
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 2 capsules orally (or via nasogastric tube) once per day starting randomization until five days after the discontinuation of the antibiotic.
  Interventions: Dietary Supplement: Placebo
- Bio K+® (Active Comparator): Bio K+® 2 capsules orally (or via nasogastric tube) once per day starting at randomization until five days after the discontinuation of the antibiotic.
  Interventions: Dietary Supplement: Bio K+® 2 capsules orally (or via nasogastric tube)

INTERVENTIONS:
Dietary Supplement: Bio K+® 2 capsules orally (or via nasogastric tube) — Bio-K+® 2 capsules orally (or via nasogastric tube) once per day starting at randomization until five days after the discontinuation of the antibiotic.
  Other Names: Bio-K+®
  Arms: Bio K+®
Dietary Supplement: Placebo — Placebo Comparator: 2 capsules orally (or via nasogastric tube) once per day starting randomization until five days after the discontinuation of the antibiotic.
  Arms: Placebo

SUMMARY:
Antibiotic-associated diarrhea (AAD) and particularly Clostridium difficile-Infection (CDI) are the most common causes of healthcare associated infectious diarrhea. In light of the results obtained in a limited number of randomized clinical trials in subjects with AAD and CDI in comparison with the widespread occurrence of these diseases, it is felt that the addition of a well-controlled clinical trial in a western environment would add value to support the use of a specific probiotic to counteract these diseases.

DETAILED DESCRIPTION:
The prevalence of Clostridium difficile infection (CDI) has been on the rise in the United States, and in fact the Centers for Disease Control and Prevention (CDC) identified CDI as one of the highest threats in its recent report on antibiotic resistance in the United States. This designation as an "urgent threat" highlights the need for immediate and aggressive action to prevent this infection.

In fact, CDI has been reported as the most commonly reported pathogen causing healthcare-associated infections (HAIs). A point prevalence survey of 183 hospitals in 10 states found that C. difficile comprised 12.1% of HAIs, surpassing Staphylococcus aureus infections.

Although most cases of CDI can be treated successfully with relatively safe and effective oral antibiotics (i.e., metronidazole or vancomycin), primary prevention of CDI is critical because up to one in five treated patients endures a relapse or reinfection, which can be difficult to treat; infected patients serve as a reservoir for ongoing transmission within facilities; implementation of contact isolation precautions for patients who have CDI can have deleterious consequences for the patient; and, CDI can result in death or severe disease including those treated by colectomy. Because CDI is spread between patients, prevention of a single case should reduce the risk of exposure for other hospital patients.

One of the main studies in this indication, being a quality improvement study conducted at Pierre Le Gardeur Hospital (PLGH) in province of Québec, Canada. Starting in 2004, 10 years of surveillance data were reported from this hospital that administers Bio-K Plus to all antibiotic users. During the 10 years of observation, 44, 835 inpatients received Bio-K+, and the CDI rate at PLGH declined from 18.0 cases per 10,000 patient-days and remained at low mean levels of 2.3 cases per 10 000 patient-days.

Additionally, 10-year data collected by the Ministry of Health in Quebec comparing the CDI rate between Quebec hospitals showed that CDI rates at PLGH were consistently and continuously lower compared with those at similar hospitals.

In conclusion, adding Bio-K Plus as a standard treatment led to a dramatic and sustained decrease in the incidence of C. difficile infections at this hospital.

ELIGIBILITY:
Inclusion Criteria

Only subjects who meet the following inclusion criteria will be eligible to participate in the study:

* Are at least 18 years old
* Able to tolerate food intake Antibiotic treatment started less than 48hrs from admission into the study
* Have an expected hospitalization period of at least three days (including subject"s stay in the emergency room)
* Speak and understand English and/or French.
* Have an expected survival greater than 60 days
* Agree to refrain from taking probiotic products (besides the study drug) during the study period Have given informed consent In addition, women of child bearing capacity who are not pregnant at the moment of screening (pregnancy test done on-site) and agree to use an acceptable form of birth control for the duration of the study (e.g. Condom, oral contraceptives, etc.) are allowed to participate.

Exclusion Criteria

Subjects who meet any of the following exclusion criteria will not be eligible to participate in the study:

* Have been diagnosed with CDI in previous sixty days
* Have taken Streptomycin, oral Vancomycin, or Metronidazole in the last 4 weeks, excluding as part of the treatment regimen triggering their inclusion into the study.
* Are currently suffering from any health condition causing immunosuppression (including haematological malignancies, lymphoma, AIDS, transplant, and hemodialysis)
* Have received more than 10 mg of prednisone per day for at least 1 month within 3 months prior to the participation to the study.
* Have active diarrhea (three or more liquid stools per 24 hour period) or non-controlled intestinal disease/colitis such as Crohn's disease, ulcerative colitis or caeliac disease Have stomas, are ostomized or are parenteral nutrition users Have already been randomized to one arm of this study
* Are known to have shown a previous reaction, including anaphylaxis, to any substance in the composition of the study products (i.e. Non-medicinal ingredients: Cellulose, hypromellose, medium chain triglycerides, sodium alginate, ascorbic acid, magnesium stearate (vegetal source), silicon dioxide and titanium dioxide
* Where receiving systemic antibiotics on admission to the hospital or who have been treated with antibiotics over the past two weeks Have lactose intolerance or milk allergy
* Have difficulties giving informed consent because of chronic mental disease, dementia
* Are not likely to comply with study requirements (provide stool for screening if diarrhea or answer to the follow up questionnaires)
* Have been known to use illicit drugs in the last two years. Have participated in another clinical study in the last 30 days
* Female subjects that are pregnant, or who intend to become pregnant or are lactating during the study period
* Female subjects of child bearing potential not currently using adequate contraception

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of Clostridium Difficile infection | 2 Years
  The primary objective of this study is evaluate the incidence risk ratio of CDI in hospitalized subjects treated with systemic antibiotics, taking oral administration of Bio-K+® in comparison with a placebo. Risk will be calculated for the period of antibiotic treatment plus 65 days.

SECONDARY OUTCOMES:
To evaluate the incidence of antibiotic associated diarrhea | 2 Years
  * To evaluate the incidence of AAD
  * To evaluate the incidence of RCDI
  * To determine the time to occurrence of the first symptoms (first liquid stool) of AAD or CDI -
  * To evaluate the impact on the duration of hospitalization
  * To evaluate the number of emergency room visits and re-hospitalizations for AAD or CDI
  * To determine the mean costs for the initial hospitalization
  * To evaluate the safety profile of Bio-K+®

CONTACTS AND LOCATIONS:
Overall Officials: Mikhael Laskine, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Serge Carriere, MD, Study Director — Bio-K+International Inc.
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada